CLINICAL TRIAL: NCT02311036
Title: Effect and Outcome Predictors on Functional Recovery After Comprehensive Rehabilitation for Post-acute Care -Cerebrovascular Diseases
Brief Title: Functional Recovery Effects on Comprehensive Rehabilitation for Post-acute Care -Cerebrovascular Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, MUJUNG KAO, Director, Taipei City Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: TCHIRB-1030404
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Cerebrovascular Diseases
Keywords: Post Acute Care(PAC); Cerebrovascular diseases
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Comorbidity_Comprehensive Rehabilitation (Other): Charlson Comorbidity Index contains 19 categories of comorbidity and predicts the ten-year mortality for a patient who may have a range of co-morbid conditions Each condition is assigned with a score of 1,2,3 or 6 depending on the risk of dying associated with this condition. For a physician, it is helpful in knowing how aggressively to treat a condition. Higher scores indicating greater comorbidity (patients with a score > 5 have essentially a 100% risk of dying at one year).
  Interventions: Other: Comprehensive Rehabilitation
- MRS_Comprehensive Rehabilitation (Other): The modified Rankin Scale (mRS) is a scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death.
  Interventions: Other: Comprehensive Rehabilitation
- MMSE_Comprehensive Rehabilitation (Other): The mini mental state examination (MMSE) is the most commonly used instrument for screening cognitive function. This examination is not suitable for making a diagnosis but can be used to indicate the presence of cognitive impairment, such as in a person with suspected dementia or following a head injury. The examination has been validated in a number of populations. Scores of 25-30 out of 30 are considered normal; the National Institute for Health and Care Excellence (NICE) classifies 21-24 as mild, 10-20 as moderate and <10 as severe impairment. The MMSE may not be an appropriate assessment if the patient has learning, linguistic/communication or other disabilities (eg, sensory impairments).
  Interventions: Other: Comprehensive Rehabilitation
- BSRS_Comprehensive Rehabilitation (Other): Brief Symptom Rating Scale is a rating scale which a clinician or researcher may use to measure psychiatric symptoms such as depression, anxiety, hallucinations and unusual behavior. Each symptom is rated 1-7 and depending on the version between a total of 18-24 symptoms are scored. The scale is the one of the oldest, widely used scales to measure psychotic symptoms and was first published in 1962.
  Interventions: Other: Comprehensive Rehabilitation

INTERVENTIONS:
Other: Comprehensive Rehabilitation — Comprehensive rehabilitation programs including PT, OT or ST will be done for two hour each every day and 5 days per week for 6-12 weeks. Initial assessment will be done within 3 days and the following assessment will be done 6 weeks or 12 weeks after rehabilitation intervention by physician and well-trained therapists.

SUMMARY:
The purpose of the study is to investigate the effects and outcome predictors on functional recovery after comprehensive rehabilitation for post-acute care -cerebrovascular diseases.

DETAILED DESCRIPTION:
The investigators will collect 165 acute stroke patients who suffer from stroke within one month and have potential of rehabilitation. The participants will be divided into mild, moderate and severe groups according to Modified Rankin Scale (MRS). The patients are admitted for 6 weeks or extend to 12 weeks if necessary after evaluation. Comprehensive rehabilitation programs including Physical Therapy (PT), Occupational Therapy (OT) or Speech Therapy (ST) will be done for two hour each every day and 5 days per week for 6-12 weeks. Initial assessment will be done within 3 days and the following assessment will be done 6 weeks or 12 weeks after rehabilitation intervention by physician and well-trained therapists. We collect basic data including sex, age, etiology of stroke, affected side, premorbid functional condition, onset time, initial function on admission, Brunnstrom stage, Charlson Comorbidity Scoring and intensity of rehabilitation. Functional assessment including: Modified Rankin Scale (MRS); Barthel Index; swallowing and feeding function, Mini Nutrition Assessment; Euro QoL-5D; Lawton-Brody IADL Scale; Berg Balance Scale (BBS); Gait speed; 6 minutes walking test; Revised Nottingham sensory assessment(RNSA); Mini-mental state examination (MMSE); Motor Activity Log(MAL); Canadian Occupational Performance Measurement(COPM); aphasia evaluation. Data analysis will be done by two-way ANOVA, paired t test, regression and multiple variant analysis.

ELIGIBILITY:
Inclusion Criteria:

* stroke patients who suffer from stroke within one month and have potential of rehabilitation
* PT, OT or ST will be done for two hour each every day and 5 days per week for 6-12 weeks.

Exclusion Criteria:

* Onset over 6 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Barthel Index improvement | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Rost NS, Smith EE, Chang Y, Snider RW, Chanderraj R, Schwab K, FitzMaurice E, Wendell L, Goldstein JN, Greenberg SM, Rosand J. Prediction of functional outcome in patients with primary intracerebral hemorrhage: the FUNC score. Stroke. 2008 Aug;39(8):2304-9. doi: 10.1161/STROKEAHA.107.512202. Epub 2008 Jun 12. PMID 18556582
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Extermann M. Measuring comorbidity in older cancer patients. Eur J Cancer. 2000 Mar;36(4):453-71. doi: 10.1016/s0959-8049(99)00319-6. PMID 10717521
- [Background] de Groot V, Beckerman H, Lankhorst GJ, Bouter LM. How to measure comorbidity. a critical review of available methods. J Clin Epidemiol. 2003 Mar;56(3):221-9. doi: 10.1016/s0895-4356(02)00585-1. PMID 12725876
- [Background] Bar B, Hemphill JC 3rd. Charlson comorbidity index adjustment in intracerebral hemorrhage. Stroke. 2011 Oct;42(10):2944-6. doi: 10.1161/STROKEAHA.111.617639. Epub 2011 Jul 28. PMID 21799172
- [Background] Goldstein LB, Samsa GP, Matchar DB, Horner RD. Charlson Index comorbidity adjustment for ischemic stroke outcome studies. Stroke. 2004 Aug;35(8):1941-5. doi: 10.1161/01.STR.0000135225.80898.1c. Epub 2004 Jul 1. PMID 15232123
- [Background] Seematter-Bagnoud L, Lecureux E, Rochat S, Monod S, Lenoble-Hoskovec C, Bula CJ. Predictors of functional recovery in patients admitted to geriatric postacute rehabilitation. Arch Phys Med Rehabil. 2013 Dec;94(12):2373-2380. doi: 10.1016/j.apmr.2013.06.024. Epub 2013 Jul 10. PMID 23850613